CLINICAL TRIAL: NCT01386242
Title: Phase II/III Study of Recombinant Anti-tumor and Anti-Virus Protein for Injection Compared With Placebo in Metastatic Colorectal Cancer After Failure of Second-Line and More Than Second-line Treatment
Brief Title: Recombinant Anti-tumor and Anti-virus Protein for Injection in Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Collaborators: Beijing Genova Biotech Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JH-RC-001; NCT02349984 (obsolete NCT alias)
Record Dates: First submitted 2011-06-27; First posted 2011-07-01 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Novaferon
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- The first group (Experimental): Recombinant anti-tumor and anti-virus protein for injection, twice per week
  Interventions: Drug: Recombinant anti-tumor and anti-virus protein for injection
- The second group (Experimental): Recombinant anti-tumor and anti-virus protein for injection, three times per week
  Interventions: Drug: Recombinant anti-tumor and anti-virus protein for injection
- Placebo group (Placebo Comparator): Saline Injection, three times per week
  Interventions: Other: Saline Injection
- The third group (Experimental): High dose of recombinant anti-tumor and anti-virus protein for injection, three times per week
  Interventions: Drug: Recombinant anti-tumor and anti-virus protein for injection

INTERVENTIONS:
Drug: Recombinant anti-tumor and anti-virus protein for injection — Recombinant anti-tumor and anti-virus protein for injection,10μg,im,twice per week for first 2 weeks, followed by 20μg, im, twice per week after 2 weeks
  Other Names: Brand name: Novaferon
  Arms: The first group
Drug: Recombinant anti-tumor and anti-virus protein for injection — Recombinant anti-tumor and anti-virus protein for injection, 10μg/1mL,im,three times per week for first 2 weeks, followed by 20μg,im, three times per week after 2 weeks.
  Other Names: Brand name: Novaferon
  Arms: The second group
Other: Saline Injection — Saline Injection, 1mL, im,three times per week
  Arms: Placebo group
Drug: Recombinant anti-tumor and anti-virus protein for injection — Recombinant anti-tumor and anti-virus protein for injection, 10μg, im, three times per week for first week, followed by 20μg for two weeks, and followed by 30μg for a week, and followed a maintenance dose of 40μg, the frequency of administration is three times per week.
  Other Names: Brand name: Novaferon
  Arms: The third group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-tumor and anti-virus protein for injection in treating patients with metastatic colorectal cancer after failure of second-line and more than second-line treatment.

DETAILED DESCRIPTION:
Explanation for study design

The trial including two stages. The first is an exploration stage to decide delivery frequency and dose of study drug. It is single-blinded, subjects will be randomly divided into 4 groups with a 2:2:2:1 ratio. Study drug given twice per week or 3 times per, dose of the drug are from 20μg to 40μg. The sample size is 105, duration is 12 to 18 months. Based on preliminary efficacy and safety, the better dosage regimen will decided for the second stage.The second stage is double-blinded,subject will be randomly divided into treatment group or placebo group with 2:1 ratio and sample size is 600.

Primary purpose

To compare overall survival between study drug and placebo groups .

Secondary purpose

1. Progression free survival were compared in both groups.
2. Disease control rate were compared in both groups.
3. Quality of life scores were compared in both groups.
4. Determine the safety and tolerance of recombinant anti-tumor and anti-virus protein for injection
5. Supplementary pharmacodynamics of recombinant anti-tumor and anti-virus protein for injection

Exploratory purpose Evaluate effects of recombinant anti-tumor and anti-virus protein for injection on the anti-tumor immunity, angiogenesis, apoptosis, cell proliferation, immune cells and cytokines levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years.
* ECOG performance status 0, 1 or 2.
* Pathologically confirmed metastatic colorectal cancer.
* Failure of Second-Line or Above Treatment, and irinotecan- and oxaliplatin--containing regimens (If recurrence and metastasis occurred within 6 months after discontinuation of adjuvant chemotherapy, the adjuvant chemotherapy is considered to be first-line treatment). more than 4 weeks before enrollment after discontinuation of chemotherapy.
* Minimum of 4 weeks since any local radiotherapy or surgery for the control of symptoms or severe complications(local radiotherapy for the control of bone metastases is not the limit)，and adequately recovered from toxicities of any prior therapy).
* At least one measurable lesion according to the RECIST criteria that has not been previously local treated. Minimum indicator lesion size as follows: greater than or equal to 10 mm measured by spiral CT or NMR.
* The organ function is normal (laboratory test results came within 1 week before administration in the absence of ongoing supportive care): ANC ≥ 1.5 x 109/L, Platelets ≥ 80 x 109/L, Hgb ≥ 8.5 g/dL, serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), and serum AST and ALT ≤ 2.5 x ULN(≤ 5 x ULN if liver metastases), serum creatinine ≤1.5 x ULN.
* Have been fully aware of the study and voluntarily signed the informed consent.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Pregnancy or breast-feeding women or women who may be pregnant were positive drug test before administration.
* Patient of child-bearing potential(male or less than 1 year postmenopausal women) were reluctant to take contraceptive measures.
* Patient who were allergic to Interferon-α or who had interferon-α antibody.
* Patients with uncontrolled central nervous system (CNS) metastases.
* Patient with any other Malignant tumors within five years (except for a complete cure of carcinoma in situ of the cervix or basal cell cancer or squamous cell skin cancer).
* Patient with Clinically uncontrolled active infection such as acute pneumonia, active hepatitis B, etc.
* Patient associated with Significant Systemic illness including, but not limited to, the following: cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, acute myocardial infarction, unstable angina, Congestive heart failure ,serious dysrhythmias, metabolic diseases, thrombosis or thromboembolic events occurred(including transient ischemic attack) in the last 6 months.
* Patient with serious autoimmune diseases in the past or at present, such as systemic lupus erythematosus, rheumatoid arthritis, thyroiditis, etc.
* Patient with ascites, pleural and pericardial effusion that cannot be controlled by drainage or symptomatic treatment.
* Investigator think Patient is not appropriate to participate in this trial for any clinical or laboratory abnormalities, or patient with any grade ≥ 2 toxicity according to NCI CTC AE 3.0 standard .
* Patient who also are accepting other systemic anti-tumor therapy (local radiotherapy for the control of bone metastases is not the limit)), in this study received 4 weeks before the start of drug treatment of other tests.
* Patient who had serious psychological or psychiatric disorder or Drug addiction or alcohol dependence.
* Patient who are estimated to be lack of compliance in this study.
* Patient with acute or subacute intestinal obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | every 8 weeks until death, the average OS is thought to be 4.5~6 months
  OS is defined as the length of time from random assignment to death or to last contact.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | every 6 weeks until disease progress, the estimate averge time is 2~3 months
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.
Quality of life (QoL) | every 2 weeks in first 4 weeks and every 4 weeks after 4 weeks, it will last to the treatment end.
  Quality of life is assessed using EORTC-C30 (the Quality of Life Questionnaire of the European Organisation for Research and Treatment of Cancer.)
Adverse Events(AEs) | from informed consent form signed to 28 days after termination of administration.
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v3.0.
pharmacodynamics | The first 2 weeks during 10ug dosage were given and the following 11weeks during 20ug dosage were given
  As the drug concentration is very low, and no commercialized kits for original drug test, So original drug will not detect. Mopterin and MxA protein (alternate index) levels in serum will be used as alternative targets for pharmacodynamic studies
Disease Control Rate | every 6 weeks until disease progression
  The disease control rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments (based on modified WHO criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Xu jianming, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Scienc
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jia R, Wang Y, Mao XY, Li SS, Xu N, Xiong JP, Shen L, Bai L, Liu W, Liu LJ, Ge FJ, Chen YL, Lin L, Xu JM. Phase II Study of Recombinant Antitumor and Antivirus Protein Injection Compared With Placebo in Metastatic Colorectal Cancer After Failure of Standard Treatment. Oncologist. 2015 Jun;20(6):619-20. doi: 10.1634/theoncologist.2014-0439. Epub 2015 Apr 29. PMID 25926350